CLINICAL TRIAL: NCT00633334
Title: Investigation of the Immune Response to Gastrointestinal Tumors and Development of Novel Biomarkers for the Presence of Gastrointestinal Cancer
Brief Title: Development of Early Detection Signs for Gastrointestinal Cancer
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Amer Zureikat, Assistant Professor, University of Pittsburgh
Other Study IDs: 02-077
Record Dates: First submitted 2008-03-03; First posted 2008-03-12 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: GI Cancer
Keywords: Cancer; GI; Tumor; Gastrointestinal; high risk
MeSH Terms: conditions — Gastrointestinal Neoplasms; Neoplasms | interventions — Biological Specimen Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — peripheral blood portions of tumor tumor draining lymph nodes
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Specimen bank — Patients will be asked to provide approximately 60-120 cc (4-8 tablespoons) of peripheral blood. Select patients who undergo surgical resection of their tumor will be asked to provide portions of the tumor and tumor draining lymph nodes for further analysis. In addition patients undergoing surgical resection may be asked to provide additional peripheral blood samples at time of routine follow-up (at least 4-6 weeks after initial blood draw and between subsequent draws).

SUMMARY:
Therapies involving the immune system have already shown great promise in early clinical trials for the treatment of renal cell carcinoma and melanoma. One of the great challenges now facing this field is to extend these findings to other cancers. Little is currently understood about the nature of the immune response to more common gastrointestinal cancers. The first goal of this proposal is to collect blood and tissue samples from patients with early or late stage gastrointestinal cancers. These samples will be evaluated to better understand the immune response to these two cancers. The second goal of this proposal is to evaluate the specimens of these patients for changes and genetic markers that correlate with the presence of cancer. The information gathered from these studies will directly enhance our ability to design, conduct and monitor novel immunotherapeutic protocols for the treatment of patients with gastrointestinal cancer.

DETAILED DESCRIPTION:
The first goal of this proposal is to collect cells from the peripheral blood, tumor draining lymph nodes and tumor infiltrating lymphocytes in patients with early or late stage gastrointestinal cancers. These samples will be evaluated in a variety of immunological assays to better understand the immune response to these two cancers. The second goal of this proposal is to evaluate using novel proteomic, cellomic, and genomic techniques the serum and peripheral blood lymphocytes of these patients for protein, cellular changes and genetic markers that correlate with the presence of cancer. The information gathered from these studies will directly enhance our ability to design, conduct and monitor novel immunotherapeutic protocols for the treatment of patients with gastrointestinal cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed GI malignancy
* suspected GI malignancy
* high risk individual as assessed by their physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects are first identified by their primary doctor/clinical team. The research project will be discussed and mutually agreed upon between the subject and his/her caregiver before the research team will contact the subject. Other subjects are referred in specifically for possible participation in a particular study which they or their physician are aware of based on publications which list clinical trials at UPMCHS.
Sampling Method: Non-Probability Sample
Enrollment: 2499 (Actual)
Dates: Start 2003-09; Primary Completion 2016-01-28 (Actual); Study Completion 2016-02-17 (Actual)

PRIMARY OUTCOMES:
The first goal of this proposal is to collect cells from the peripheral blood, tumor draining lymph nodes and tumor infiltrating lymphocytes in patients with early or late stage gastrointestinal cancers. | 1 N/A

SECONDARY OUTCOMES:
The second goal is to evaluate using novel proteomic, CellomicTM, and genomic techniques the serum and peripheral blood lymphocytes of these patients for protein, cellular changes and genetic markers that correlate with the presence of cancer. | 1 N/A

CONTACTS AND LOCATIONS:
Overall Officials: Herber J. Zeh, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States